CLINICAL TRIAL: NCT05601700
Title: Letrozole for Estrogen/Progesterone Receptor Positive Low-grade Serous Epithelial Ovarian Cancer: a Randomized Phase III Trial (LEPRE Trial)
Brief Title: Letrozole for Estrogen/Progesterone Receptor Positive Low-grade Serous Epithelial Ovarian Cancer (LEPRE Trial)
Acronym: LEPRE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other); Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Andrea DeCensi, Medical Oncology Director, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10UCS2018; 2020-003066-39 (EudraCT Number)
Record Dates: First submitted 2022-10-21; First posted 2022-11-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Ovarian Epithelial; Low Grade Serous Adenocarcinoma of Ovary
Keywords: Estrogen/progesteron receptor positive tumor; Letrozole; Aromatase Inhibitors
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Letrozole; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Letrozole 2.5 mg daily, per os, until progression or up to 60 months, whichever comes first
  Interventions: Drug: Letrozole tablets
- Control arm (Active Comparator): Carboplatin AUC 5 + Paclitaxel 175 mg/mq, IV, on day 1 every 21 days, for 6-8 cycles.
  Interventions: Drug: carboplatin AUC 5 and paclitaxel 175 mg/m2

INTERVENTIONS:
Drug: Letrozole tablets — ATC: L02BG04
  Arms: Experimental arm
Drug: carboplatin AUC 5 and paclitaxel 175 mg/m2 — ATC: L01XA02 and ATC: L01CD01 respectively
  Arms: Control arm

SUMMARY:
This is an Italian, multicenter, randomized, open-label phase III trial which will evaluate if Letrozole is superior to standard adjuvant chemotherapy in patients with hormone receptor positive low-grade serous epithelial carcinoma of the ovary (LGSCO).

The hypothesis is that letrozole will significantly prolong median progression free survival (PFS) compared with the standard chemotherapy treatment, namely carboplatin AUC 5 and paclitaxel 175 mg/m2.

DETAILED DESCRIPTION:
Primary objective:

To determine if letrozole is superior to standard chemotherapy in terms of progression-free survival (PFS) in the first line treatment of patients with advanced low-grade serous epithelial ovarian carcinoma positive for estrogen and/or progesterone receptors.

Secondary objectives:

* to evaluate the response of tumor to letrozole compared with standard chemotherapy in terms of objective response rate (ORR);
* to test the predictive effect of ER and PgR on response to letrozole in terms of PFS and ORR;
* to evaluate the possible negative association between the effect of letrozole, in terms of PFS and ORR, and the proliferative index Ki67;
* to evaluate the impact of letrozole compared with the impact of standard chemotherapy on patients' health related quality of life evaluated by Menopausal Quality of Life Questionnaire (MENQOL);
* to evaluate the impact of letrozole compared with standard chemotherapy on patients' musculoskeletal pain evaluated by Brief Pain Inventory - Short Form (BPISF);
* to evaluate the effect on overall survival (OS). As most patients will recur and will be switched to chemotherapy and vice versa, OS is not expected to be significantly different;
* to evaluate the safety of letrozole compared with standard chemotherapy according to CTCAE v 5.0.

Translational objectives:

* to characterize the mutational profile and gene expression of the disease by NGS (next-generation sequencing) methodology on tissue samples;
* to evaluate the circulating tumor DNA (ctDNA) on liquid biopsies as a tool to monitor the disease response.

ELIGIBILITY:
Inclusion Criteria:

I - 1. Age ≥ 18 years. I - 2. Newly diagnosed, low-grade serous carcinoma of the ovary including cancer of fallopian tube and peritoneum (invasive micropapillary serous carcinoma or invasive grade 1 serous carcinoma). This is to be confirmed via nuclear p53 immunohistochemistry testing by a central pathology review performed at the Coordinating Centre.

I - 3. Immunohistochemically determined positivity (≥ 10%) for ER and/or PgR expression. This is to be confirmed by centralized review.

I - 4. Patients must have undergone an upfront surgery with maximal cytoreductive effort, with either optimal or suboptimal residual disease status.

I - 5. Stage III-IV according to 2018 FIGO classification. For proper staging:

* Patients must have undergone contrast-enhanced CT-scan of the chest, abdomen and pelvis within 28 days prior to randomization. If CT-scan is not recommended (e.g. for allergy to contrast agent) MRI or 18F-FDG PET/CT-scan are allowed.
* The imaging evaluation must be accompanied by an anamnestic and physical examination within 14 days prior to randomization.

I - 6. Postmenopausal, defined as any of the following criteria:

* Patients who underwent bilateral salpingo-oophorectomy;
* Monolateral salpingo-oophorectomy, amenorrhea for 12 or more consecutive months and age ≥60 years;
* Monolateral salpingo-oophorectomy, amenorrhea for 12 or more consecutive months, age <60 years and FSH and serum estradiol levels within the laboratory's reference ranges for post-menopausal women.

I - 7. Randomization must take place within 60 days of primary cytoreductive surgery.

I - 8. Eastern Cooperative Oncology Group - performance status (ECOG-PS) 0-1.

I - 9. To be able to take oral medications.

I - 10. Adequate bone marrow, hepatic and renal functions as defined below:

* Absolute neutrophil count (ANC) ≥ 1500/mm3
* Platelets ≥ 100,000/mm3
* Hemoglobin ≥ 10.0 g/dL
* Total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN)
* ALT and AST ≤ 3.0 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Albumin ≥ 2.8 g/dL
* Serum creatinine ≤ 1.5 x ULN.

I - 11. Written informed consent obtained prior to any study-specific procedure.

Exclusion Criteria:

E - 1. Other malignancy within the last 5 years, except for non-melanoma skin cancer adequately treated.

E - 2. Neoadjuvant chemotherapy or radiotherapy for the treatment of this disease.

E - 3. Previous hormonal therapy for the treatment of this disease.

E - 4. Known hypersensitivity to letrozole or known hypersensitivity/intolerance to carboplatin/paclitaxel therapy.

E - 5. Active or uncontrolled systemic infection.

E - 6. Known central nervous system metastases.

E - 7. Severe cardiac disease, such as myocardial infarction or unstable angina within 6 months prior to randomization.

E - 8. New York Heart Association (NYHA) Class III or greater congestive heart failure.

E - 9. Neuropathy grade 2 or higher.

E - 10. History of fractures of the spine or femur not properly treated.

E - 11. Known osteoporosis (dual-energy x-ray absorptiometry (DEXA) of the femoral neck T score of -2.5 or lower) not adequately treated with bisphosphonates or RANKL inhibitors.

E - 12. Concomitant use of inducers of CYP3A4 (e.g. phenytoin, rifampicin, carbamazepine, phenobarbital, and St. John's Wort) which may reduce exposure to letrozole. Concomitant use of medicinal products with a narrow therapeutic index that are substrates for CYP2C19 (e.g. phenytoin, clopidrogel) that may have their systemic serum concentrations altered by letrozole.

E - 13. Concurrent severe medical problems or any condition that would significantly limit full compliance with the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2029-09-22 (Estimated); Study Completion 2029-09-22 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 54 months up to 84 months
  the time from the date of randomization to the date of local or regional relapse, distant metastasis, or death from any cause, whichever comes first. Patients not recurred, not progressed or not died while on study or patients lost to f-up will be censored at their last disease assessment date.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 54 months up to 84 months
  the percentage of patients with an objective response, i.e. patients who will experience a complete response (CR), or a partial response (PR) as determined by RECIST 1.1. Each patient will be assigned the best response ever recorded during the trial.
Predictive effect of ER and PgR (% expression) on response to letrozole in terms of PFS and ORR | 54 months up to 84 months
  the time from the date of randomization to the date of local or regional relapse, distant metastasis, or death from any cause, whichever comes first according to ER and PgR % expression.
Clinical Benefit (CB) | 54 months up to 84 months
  the percentage of patients who will experience a CR or PR or stable disease (SD). Each patient will be assigned the best response ever recorded during the trial.
Overall survival (OS) | 54 months up to 84 months
  the time from the date of randomization to the date of death from any cause. Patients not reported as having died at the end of the study will be censored at the date they were last known to be alive.
Safety (Adverse Events) | 54 months up to 84 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE

OTHER OUTCOMES:
Translational Objective 1 | 54 months up to 84 months
  mutational and gene expression profile of the disease by means of NGS based methodology on tissue
Translational Objective 2 | 54 months up to 84 months
  PFS, OS and ORR according to androgen receptor (AR) expression
Translational Objective 3 | 54 months up to 84 months
  PFS, OS and ORR according to circulating tumor DNA (ctDNA) on liquid biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Andrea DeCensi, MD, Principal Investigator — E.O.Ospedali Galliera
Locations (19):
- Italy (19):
  - Ospedale San Donato, Arezzo, AR
  - Ospedale degli Infermi, Ponderano, BI
  - Ospedale San Martino, Belluno, BL
  - Fondazione Poliambulanza, Brescia, BS
  - ASST degli Spedali Civili di Brescia, Brescia, BS
  - Ospedale Sant'Anna, Como, CO
  - IRST, Meldola, FC
  - AOU Ferrara, Ferrara, FE
  - Medical Oncology Division, Ente Ospedaliero Ospedali Galliera, Genova, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - IEO, Milan, MI
  - IRCCS Istituto Oncologico Veneto, Padua, PD
  - IFO Regina Elena, Roma, RM
  - Policlinico Umberto I, Roma, RM
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - IRCCS Istituto Oncologico Veneto, Castelfranco Veneto, TV
  - Ospedale Ca' Foncello, Treviso, TV
  - Ospedale Del Ponte, Varese, VA
  - AUSL Romagna, Rimini

REFERENCES:
- [Derived] Carbone A, Biagioli E, Salutari V, Lorusso D, Provinciali N, Bocciolone L, Artioli G, Abeni C, Colombo N, De Giorgi U, Guarneri V, Cassani C, Scarfone G, Zavallone L, Donadello N, Donato VD, Giordano M, Scelzi E, Tognon G, Petrella MC, D'Incalci M, Marchini S, Dang HT, Alvisi MF, Corradengo D, Buttiron Webber T, Paleari L, Briata IM, Rutigliani M, Oliva M, Rulli E, DeCensi A. Letrozole for hormone receptor-positive low-grade ovarian cancer: Preliminary toxicity results of a phase III trial. Tumori. 2025 Dec 14:3008916251395596. doi: 10.1177/03008916251395596. Online ahead of print. PMID 41392465